CLINICAL TRIAL: NCT05892445
Title: Impact of Aversive Visual Health Warnings on E-Cigarette Cessation Intentions and Behaviors Among Young Adults
Brief Title: Impact of Aversive Warnings on E-Cigarette Cessation
Status: Not yet recruiting | Phase: Phase 3 | Type: Interventional
Sponsor: University of California, San Diego (Other)
Responsible Party: Principal Investigator, Raphael Cuomo, Assistant Professor, University of California, San Diego
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Other
Other Study IDs: 1422045
Record Dates: First submitted 2023-05-26; First posted 2023-06-07 (Actual); Last update posted 2024-06-05 (Actual); Status verified 2024-06

CONDITIONS: E Cigarette Use
MeSH Terms: conditions — Vaping

STUDY DESIGN:
Who Masked: Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Aversive Visual Health Warnings (Experimental): Study subjects in this arm will be exposed to experimental aversive visual health warnings depicting risks and adverse effects of e-cigarette use. They will answer survey questions about e-cigarette perceptions before and after exposure to health warnings.
  Interventions: Behavioral: Graphic Warning Labels
- No Warnings (No Intervention): Study subjects in this arm will answer the same survey questions about e-cigarette perceptions as those in the experimental arm, but they will not be shown aversive visual health warnings.

INTERVENTIONS:
Behavioral: Graphic Warning Labels — Based on a thorough review of the literature on e-cigarette risks and adverse effects, a graphic designer will be contracted to create ten experimental aversive health warnings related to e-cigarettes. These warnings will be exported as high-quality images and shown to participants in the intervention group prior to questions that obtain data on the primary endpoint.
  Arms: Aversive Visual Health Warnings

SUMMARY:
This project aims to evaluate the effectiveness of aversive visual health warnings on e-cigarette cessation among young adults through a randomized controlled trial, as e-cigarette use among this population has been steadily increasing, posing significant public health concerns. While traditional tobacco products have long featured health warnings, e-cigarettes lack similarly aversive visual warnings, and this study seeks to inform the development of targeted e-cigarette cessation strategies and contribute to a deeper understanding of how visual health warnings can be utilized to reduce e-cigarette use and ultimately improve public health. The project has three main aims, which include a rigorous assessment of the academic literature on e-cigarette risks and adverse effects to develop evidence-based mock visual health warnings for e-cigarettes; assessing the effectiveness of aversive visual health warnings in increasing intent to cessate e-cigarettes, with a particular focus on individuals who have experienced adverse events; and examining the long-term impacts of visual health warnings on e-cigarette cessation. This study will also investigate the underlying mechanisms that may explain the relationship of the intervention on cessation. To generate visual warnings, the research team will conduct a thorough review of the scientific literature on e-cigarette risks and adverse effects and collaborate with a graphic designer. Experimental warnings will be annotated and categorized in order to understand the influence of different imagery on variations in participant response. The study will be conducted as a randomized controlled trial, recruiting participants through market research firms that will distribute an online survey to their panels of e-cigarette users. Participants will be eligible for inclusion if they are 18-29 years old and currently use e-cigarettes at least once per week. A quota will be included to ensure sufficient responses from individuals who have experienced at least one adverse event related to e-cigarette use in the past 12 months. The intervention group will be exposed to a series of aversive visual health warnings about the potential health risks of e-cigarette use, delivered through the online survey platform, while the control group will not receive any intervention and will complete the same survey as the intervention group. Data will be analyzed using appropriate statistical techniques, including logistic regression and mediation/moderation analysis, to assess the effectiveness of the aversive visual health warnings in reducing e-cigarette use and the moderating effects of prior adverse event experience. Participants will be contacted for follow-up assessments at 3-months post-intervention to investigate the impact of aversive visual health warnings on e-cigarette cessation among young adults, including the moderating effects of prior adverse event experience, and assess the underlying mechanisms that may explain the relationship between the intervention and e-cigarette cessation.

ELIGIBILITY:
* Age 18-29 years
* Basic understanding of English
* Not institutionalized
* Currently use e-cigarettes at least once per week

Ages: 18 Years to 29 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 1000 (Estimated)
Dates: Start 2025-05-01 (Estimated); Primary Completion 2025-09-30 (Estimated); Study Completion 2025-09-30 (Estimated)

PRIMARY OUTCOMES:
Intent to Cessate Use of E-Cigarettes | Immediately after exposure to intervention
  Every participant will take a survey with a question that asks about willingness to cease e-cigarettes using the seven-point Motivation To Stop Scale, adapted for e-cigarettes, in order to assess the influence of the intervention.

SECONDARY OUTCOMES:
E-Cigarette Cessation Attempt | Six months after exposure to intervention
  Participants completing the first survey will be recontacted six months after their completion date to complete a second survey. This survey will ask whether the participant has made an attempt to quit using e-cigarettes, as well as the approximate date of the quit attempt.

IPD SHARING:
Plan to Share IPD: Yes
The project will generate survey data collected from 1000 young adult e-cigarette users, along with follow-up data from the same participants at 3 months post-intervention. The anonymized survey data and follow-up data will be preserved and shared to facilitate further analysis and replication of the study. The data will include demographics, e-cigarette use patterns, intentions to quit, perceived risk and harm, exposure to health warnings, and experiences with adverse events.
Supporting Information: Analytic Code
Time Frame: The dataset will be made available within 12 months of project completion (following publication of primary findings) and will be maintained for a minimum of 10 years.
Access Criteria: Users will be required to register and agree to use the data for research purposes only.